CLINICAL TRIAL: NCT06501937
Title: The Impact of Healthy Lifestyle Imagery Alongside E-cigarettes in Social Media Influencer Marketing on Perceptions of E-cigarettes Among Adolescents: a Survey-based Experiment
Brief Title: Influencer Marketing: a Survey-based Experiment Among Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Jennifer Unger, Professor, University of Southern California
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: UP-21-00352
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Intervention Model Description: Videos featuring influencers promoting e-cigarettes alongside healthy lifestyle activities
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Videos featuring influencers promoting e-cigarettes alongside healthy lifestyle activities
  Interventions: Other: Influencer marketing
- Control group (Active Comparator): Videos featuring influencers promoting e-cigarettes alone
  Interventions: Other: Influencer marketing

INTERVENTIONS:
Other: Influencer marketing — Participants watched online survey-imbedded promotional videos featuring influencers

SUMMARY:
Adolescents (N = 664) participated in the online survey-based experiment. They were randomly shown 10 videos, featuring influencers promoting e-cigarettes alongside healthy lifestyle activities (experimental group), or e-cigarette promotion alone (control). After watching each video, participants rated perceptions of influencer credibility (i.e., honesty, trustworthiness, knowledge) on the scale of 0 (e.g., dishonest) to 100 (honest).

Among all participants, harm perceptions and appeal of e-cigarettes was assessed. Susceptibility to use e-cigarettes was assessed among never users of e-cigarettes. These outcomes were then compared among participants who perceived influencers as credible and those who perceived influencers as non-credible.

DETAILED DESCRIPTION:
Adolescents (13-17 years of age) living in California were recruited by Qualtrics marketing research panel to participate in a survey on tobacco-related attitudes and behaviors. Qualtrics, a research panel agency, has been used in prior research to survey adolescents about their tobacco-related attitudes and behaviors. Participants were provided with a survey URL link. After completing informed consent, participants completed the survey online. The study was approved by the University of Southern California Institutional Review Board (UP-21-00352). Respondents were randomly assigned to watch 10 10-second long TikTok videos in either experimental (influencers promoting e-cigarettes alongside healthy lifestyle activities) or control group (influencers promoting e-cigarettes alone).

ELIGIBILITY:
Inclusion Criteria:

* 13-17 years of age,
* English fluency,
* Current California resident.

Exclusion Criteria:

Not meeting these criteria:

* 13-17 years of age,
* English fluency,
* Current California resident.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 664 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Harm perceptions of e-cigarettes | one-time assessment after the experimental exposure (immediately post-treatment)
  Responses to two questions adapted from PATH, "Based on the videos you just watched, do you think using e-cigarettes for vaping nicotine is harmful to your health?" "Based on the videos you just watched, do you think people harm themselves when they use e-cigarettes for vaping nicotine?" Outcome was assessed on the 0 (Not harmful at all) - 100 (Very harmful) scale. Since the items were closely related (α=0.87), they were combined (by summing all the non-missing values of the items) into one variable.
Perceived appeal of e-cigarettes | one-time assessment after the experimental exposure (immediately post-treatment)
  Responses to the following questions: using e-cigarette is:
  * not cool/cool,
  * unattractive/attractive,
  * boring/fun were assessed on the 7-point semantic differential scale with the word pairs anchored at each end. The scale was adapted from prior research. The items were combined (by summing all the non-missing values of the items) into one variable (α=0.93).
Susceptibility to use e-cigarettes | one-time assessment after the experimental exposure (immediately post-treatment)
  Susceptibility to use e-cigarettes was measured (among never-users of e-cigarettes), using the validated three-item scale adapted from PATH, and combined into one variable (α=0.93). Consistent with prior research, the measure was dichotomized with responses "definitely not" to all items being coded as "not susceptible" and responses "probably not," "probably yes", or "definitely yes" being coded as "susceptible."
Perceptions of influencer credibility | assessed 10 times immediately after each video
  Perceptions of influencer credibility (i.e., honesty, trustworthiness, knowledge) were assessed using a 0 (e.g., dishonest) -100 (e.g., honest) scale that has been validated in prior research.

CONTACTS AND LOCATIONS:
Locations (1):
- Online survey, Qualtrics, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No
de-identified data will be publicly available on GitHub repository if a manuscript related to this study is accepted for publication